CLINICAL TRIAL: NCT04608682
Title: Effect of Intraoperative Muscle Relaxation Reversal on the Success Rate of Motor Evoked Potential Recording
Brief Title: Effect of Muscle Relaxation Reversal on the Success Rate of Motor Evoked Potential Recording
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WJP20201030
Record Dates: First submitted 2020-10-25; First posted 2020-10-29 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Sugammadex; Motor Evoked Potentials
MeSH Terms: interventions — Sugammadex; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugammadex group (Experimental)
  Interventions: Drug: Sugammadex
- control group (Sham Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Sugammadex — The muscle relaxant infusion will be discontinued and a bolus of sugammadex (2mg/kg) will be given while performing TceMEPs.
  Arms: Sugammadex group
Drug: Saline — The muscle relaxant infusion will be discontinued and 2ml saline will be infused, TceMEPs monitoring will be performed 5 minutes later.
  Arms: control group

SUMMARY:
Transcranial motor evoked potential (TcMEP) monitoring is conventionally performed during surgery without or with minimal neuromuscular blockade (NMB) because of its potential interference with signal interpretation.The feasibility of TcMEP interpretation was assessed during partial NMB in adult neurosurgical patients. However, partial NMB may interfere record of TcMEP monitoring. Sugammadex is the first highly selective antagonist that can reverse NMB. This study aims to evaluate the success rate of intraoperative muscle relax reversal by sugammadex on intraoperative TceMEP recording.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 65 years old
* American Society of Anesthesiologists (ASA) physical status I to II

Exclusion Criteria:

* BMI ≥35 kg/m-2
* History of epilepsy or use of antiepileptic drugs
* Personal history or family history of malignant hyperthermia
* Allergies to sugammadex; NMBs or other medication(s) used during general anesthesia
* Hemoglobin <110 g/L
* TceMEP stimulation or recorded site infection
* Preoperative neurological dysfunction in both upper extremities
* Cardiac pacemaker
* Pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
The success rate of TceMEPs | 5 minutes after first performing of TceMEPs
  The success rate of Transcranial motor evoked potentials monitoring（TceMEPs）

SECONDARY OUTCOMES:
Mean value of amplitudes of TceMEPs | 5, 10, 20, 30 and 60 minutes after first performing of TceMEPs
  Mean value of amplitudes of Transcranial motor evoked potentials monitoring（TceMEPs）in the abductor pollicis brevis muscles of both upper extremities
Mean value of latencies of TceMEPs | 5, 10, 20, 30 and 60 minutes after first performing of TceMEPs.
  Mean value of latencies of Transcranial motor evoked potentials monitoring（TceMEPs） in the abductor pollicis brevis muscles of both upper extremities
Thresholds of TceMEPs | 5 minutes after first performing of TceMEPs
  The thresholds that are required to obtain a dependable Transcranial motor evoked potentials monitoring（TceMEPs） response.
respiratory pressure | during the surgery
  Peak respiratory pressures
Adverse effects of sugammadex | during the surgery
  Adverse effects of sugammadex such as anaphylaxis (including flushing, oedema, tachycardia and bronchospasm), arrhythmias (heart rate lower than 60bpm), postprocedural pain, nausea and vomiting, fever (body temperature more than 37.3℃ ), and diarrhea, etc
Incidence of body movement | during the surgery
  Incidence of body movement classified as either nociception-induced movement (defined as "coughing" or reflexive limb movement temporally related to MEP stimulation) or excessive field movement (defined as grossly visible movement as determined by surgical and anaesthesia teams).
Recurrence of neuromuscular blockade | time of extubation
  Recurrence of neuromuscular blockade defined as TOFr < 0.9

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months after the study is finished
Access Criteria: principal investigator

REFERENCES:
- [Derived] Jian M, Liu H, Liang F, Ma B, Wang L, Zhou Y, Qiao H, Han R, Wang C. Effect of intraoperative muscle relaxation reversal on the success rate of motor evoked potential recording in patients undergoing spinal surgery: a randomized controlled trial. BMC Anesthesiol. 2023 Aug 25;23(1):290. doi: 10.1186/s12871-023-02211-z. PMID 37626303
- [Derived] Jian M, Ma B, Liu H, Wang C, Liang F, Zhou Y, Qiao H, Han R. Effect of intraoperative muscle relaxation reversal on the success rate of motor-evoked potential recording in patients undergoing spinal surgery: study protocol for a randomised controlled trial. BMJ Open. 2022 May 2;12(5):e056571. doi: 10.1136/bmjopen-2021-056571. PMID 35501072